CLINICAL TRIAL: NCT01077154
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase 3 Study of Denosumab as Adjuvant Treatment for Women With Early-Stage Breast Cancer at High Risk of Recurrence (D-CARE)
Brief Title: Study of Denosumab as Adjuvant Treatment for Women With High Risk Early Breast Cancer Receiving Neoadjuvant or Adjuvant Therapy (D-CARE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated: Amgen decision following Primary Analysis. Not due to safety reason
Sponsor: Amgen (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060359; 2009-011299-32 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-26 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Early Stage Breast Cancer; Bone Metastasis; Adjuvant treatment; Neoadjuvant treatment; Denosumab; Stage II breast cancer; Stage III breast cancer; Stage IIA breast cancer; Stage IIB breast cancer; Stage IIIA breast cancer; Stage IIIB breast cancer; Stage IIIC breast cancer; Early breast cancer; Breast Tumors; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections once every 4 weeks for 6 months followed by placebo subcutaneous injections once every 3 months for 4.5 years.
  Interventions: Drug: Placebo
- Denosumab (Experimental): Participants received denosumab 120 mg subcutaneous injections once every 4 weeks for 6 months followed by denosumab 120 mg subcutaneous injections once every 3 months for 4.5 years.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Placebo — Administered subcutaneously for up to 5 years
  Arms: Placebo
Drug: Denosumab — Administered subcutaneously for up to 5 years
  Other Names: XGEVA®
  Arms: Denosumab

SUMMARY:
This randomized phase 3 trial is studying the effect of denosumab to see if it can prevent disease recurrence in the bone or in any other part of the body, when it is given as adjuvant therapy for women with early-stage breast cancer, who are at high risk of disease recurrence.

DETAILED DESCRIPTION:
Eligible participants were randomized in a 1:1 ratio to receive denosumab 120 mg or placebo subcutaneously (SC) for up to 5 years. Randomization was stratified based on:

1. Breast cancer therapy/lymph node (LN) status: neoadjuvant therapy/any LN status versus adjuvant therapy/LN negative (based on axillary LN dissection, or based on sentinel node status) versus adjuvant therapy/LN positive
2. Hormone receptor (estrogen receptor [ER]/progesterone receptor [PR]) status: ER and/or PR positive versus ER and PR negative
3. Human epidermal growth factor receptor 2 (HER-2) status: HER-2 positive versus HER-2 negative
4. Age: < 50 years versus ≥ 50 years
5. Geographic Region: Japan versus Other regions.

The primary analysis was conducted after all enrolled participants had the opportunity to complete 5 years of treatment from study day 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, American Joint Committee on Cancer (AJCC) stage II or III breast cancer
* High risk of breast cancer recurrence, defined as documented evidence of one or more of the following criteria:

  i) Biopsy evidence of breast cancer in regional lymph node(s) (LN) (node-positive disease); Nodal micrometastases only are not considered node positive ii) Tumor size > 5 cm (T3) or locally advanced disease (T4)
* Documented pathological evaluation of the breast cancer for hormone receptor (estrogen receptor [ER] and progesterone receptor [PR]) status and HER-2 status
* Subjects must be receiving or be scheduled to receive standard of care systemic adjuvant or neoadjuvant chemotherapy and/or endocrine therapy and/or HER-2 targeted therapy
* For subjects receiving adjuvant therapy only:
* subjects must have undergone complete resection of the primary tumor with clean surgical margins, or subjects must have undergone resection of the primary tumor and be scheduled for further treatment of the primary tumor with curative intent. Definitive treatment must be planned to be completed within approximately 9 months of randomization
* Time between definitive surgery and randomization must be ≤ 12 weeks. Definitive surgery may include secondary interventions (e.g. to clear inadequate surgical margins)
* Subjects with node positive disease must have undergone treatment of axillary LN with curative intent, or subjects must be scheduled for further treatment of regional lymph nodes with curative intent. Definitive treatment must be planned to be completed within approximately 9 months of randomization
* Subjects must not have received prior neoadjuvant treatment. Endocrine treatment for less than 30 days prior to surgery is not considered prior neoadjuvant treatment
* For subjects receiving neoadjuvant therapy only:
* Time between start of neoadjuvant treatment and randomization must be ≤ 8 weeks and subjects must be scheduled to undergo definitive treatment (including surgery and/or radiotherapy) with curative intent within approximately 9 months of starting neoadjuvant treatment
* Female subjects with age ≥ 18 years
* Subjects with reproductive potential must have a negative pregnancy test within 14 days before randomization
* Serum calcium or albumin-adjusted serum calcium ≥ 2.0 mmol/L (8.0 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Written informed consent before any study-specific procedure is performed

Exclusion Criteria:

* Prior or current evidence of any metastatic involvement of any distant site
* History of breast cancer (other than ductal carcinoma in situ [DCIS] or lobular carcinoma in situ [LCIS]) prior to the current diagnosis
* Osteoporosis requiring treatment at the time of randomization or treatment considered likely to become necessary within the subsequent six months
* Any prior or synchronous malignancy (other than breast cancer), except i) Malignancy treated with curative intent and with no evidence of disease for ≥ 5 years prior to enrollment and considered to be at low risk for recurrence by the treating physician ii) Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Active infection with Hepatitis B virus or Hepatitis C virus
* Known infection with human immunodeficiency virus (HIV)
* Prior history or current evidence of osteomyelitis/osteonecrosis of the jaw
* Active dental or jaw condition which requires oral surgery
* Planned invasive dental procedure for the course of the study
* Non-healed dental or oral surgery
* Use of oral bisphosphonates within the past 1 year
* Prior or current IV bisphosphonate administration
* Prior administration of denosumab
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or investigational drug study(s), or subject is receiving other investigational agent(s)
* Subject is pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment.
* Subject is of child bearing potential and is not willing to use, in combination with her partner, 2 highly effective methods of contraception or abstinence during treatment and for 5 months after the end of treatment
* Subject has known sensitivity to any of the products to be administered during the study (e.g., mammalian derived products, calcium, or vitamin D)
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* Any major medical or psychiatric disorder that in the opinion of the investigator prevent the subject from completing the study or interfere with the interpretation of the study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4509 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (390):
- United States (84):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Campbell, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, La Verne, California
  - Research Site, Lancaster, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Redondo Beach, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Maria, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Grand Junction, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Athens, Georgia
  - Research Site, Niles, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Paducah, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Danvers, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Denville, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, East Setauket, New York
  - Research Site, New York, New York
  - Research Site, Nyack, New York
  - Research Site, Asheville, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Garland, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Richlands, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Argentina (5):
  - Research Site, Quilmes, Buenos Aires
  - Research Site, San Martín, Buenos Aires
  - Research Site, Neuquén, NeuquÃ©n
  - Research Site, Provincia de Santa Fe, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Australia (20):
  - Research Site, Camperdown, New South Wales
  - Research Site, Caringbah, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Bedford Park, South Australia
  - Research Site, Bentleigh East, Victoria
  - Research Site, East Melbourne, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Frankston, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Richmond, Victoria
  - Research Site, Ringwood East, Victoria
  - Research Site, Warrnambool, Victoria
  - Research Site, Wodonga, Victoria
  - Research Site, Perth, Western Australia
  - Research Site, Subiaco, Western Australia
- Belgium (18):
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, LiÃ¨ge
  - Research Site, Libramont
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Ottignies
  - Research Site, Sint-Niklaas
  - Research Site, Tournai
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Brazil (9):
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Curitiba, ParanÃ¡
  - Research Site, Londrina, ParanÃ¡
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, ItajaÃ-, Santa Catarina
  - Research Site, Barretos, SÃ£o Paulo
  - Research Site, Santo André, SÃ£o Paulo
  - Research Site, São Paulo, SÃ£o Paulo
  - Research Site, SÃ£o Paulo, SÃ£o Paulo
- Bulgaria (6):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (19):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Sydney, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (3):
  - Research Site, Temuco, CautÃ-n
  - Research Site, Viña del Mar, ValparaÃ-so
  - Research Site, Santiago
- Czechia (6):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Denmark (4):
  - Research Site, Ã…rhus C
  - Research Site, Herning
  - Research Site, Vejle
  - Research Site, Viborg
- France (14):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, HyÃ¨res
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Monaco
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Bottrop
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Kiel
  - Research Site, Koblenz
  - Research Site, Mannheim
  - Research Site, MÃ¼nchen
  - Research Site, Recklinghausen
  - Research Site, Rostock
  - Research Site, TÃ¼bingen
  - Research Site, Trier
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- India (11):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Ahilyanagar, Maharashtra
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Miraj, Maharashtra
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
- Ireland (4):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Limerick
  - Research Site, Waterford
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Poria Eylit
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (11):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Meldola FC
  - Research Site, Milan
  - Research Site, Monza (MB)
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, San Giovanni Rotondo FG
  - Research Site, Treviglio (BG)
  - Research Site, Varese
- Japan (23):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Kure-shi, Hiroshima
  - Research Site, Akashi-shi, Hyōgo
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Isehara-shi, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Miyazaki, Miyazaki
  - Research Site, Niigata, Niigata
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Hidaka-Shi, Saitama
  - Research Site, Kitaadachi-gun, Saitama
  - Research Site, Suntou-gun, Shizuoka
  - Research Site, Shimotsuke-shi, Tochigi
  - Research Site, Utsunomiya, Tochigi
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Tokyo
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Liepāja
  - Research Site, Riga
- Malaysia (3):
  - Research Site, Kota Bharu, Kelantan
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Subang Jaya, Selangor (incl. Putrajaya)
- Mexico (10):
  - Research Site, León, Guanajuato
  - Research Site, Pachuca, Hidalgo
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo LeÃ³n
  - Research Site, Querétaro, QuerÃ©taro
  - Research Site, San Luis Potosí City, San Luis PotosÃ-
  - Research Site, Colima
  - Research Site, Distrito Federal
  - Research Site, Durango
  - Research Site, Toluca
- Netherlands (15):
  - Research Site, Amsterdam
  - Research Site, Bergen op Zoom
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Dordrecht
  - Research Site, Hoofddorp
  - Research Site, Leiden
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sittard-Geleen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Venlo
- Research Site, Lima, Peru
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Metro Manila
  - Research Site, Quezon City
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Szczecin
- Portugal (3):
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Santa Maria da Feira
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Sibiu
  - Research Site, Suceava
  - Research Site, Timișoara
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niš
- Slovakia (7):
  - Research Site, Bardejov
  - Research Site, Košice
  - Research Site, Michalovce
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Spišská Nová Ves
  - Research Site, Trebišov
- Slovenia (2):
  - Research Site, Ljublijana
  - Research Site, Maribor
- South Africa (6):
  - Research Site, Groenkloof, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town
  - Research Site, Pietermaritzburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (3):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (17):
  - Research Site, CÃ³rdoba, AndalucÃ-a
  - Research Site, CÃ¡diz, AndalucÃ-a
  - Research Site, JaÃ©n, AndalucÃ-a
  - Research Site, MÃ¡laga, AndalucÃ-a
  - Research Site, Seville, AndalucÃ-a
  - Research Site, Zaragoza, AragÃ³n
  - Research Site, Santander, Cantabria
  - Research Site, Badalona, CataluÃ±a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Girona, CataluÃ±a
  - Research Site, Lleida, CataluÃ±a
  - Research Site, Sabadell, CataluÃ±a
  - Research Site, A CoruÃ±a, Galicia
  - Research Site, AlcorcÃ³n, Madrid
  - Research Site, Elche, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Taiwan (4):
  - Research Site, Putzu City, Chiayi
  - Research Site, Keelung, Keelung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Ä°zmir
  - Research Site, Bornova-Izmir
- United Kingdom (17):
  - Research Site, Bebington
  - Research Site, Birmingham
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Dorset
  - Research Site, Guildford
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, Peterborough
  - Research Site, Plymouth
  - Research Site, Poole
  - Research Site, Portsmouth
  - Research Site, Sheffield
  - Research Site, Truro

REFERENCES:
- [Background] Coleman R, Finkelstein DM, Barrios C, Martin M, Iwata H, Hegg R, Glaspy J, Perianez AM, Tonkin K, Deleu I, Sohn J, Crown J, Delaloge S, Dai T, Zhou Y, Jandial D, Chan A. Adjuvant denosumab in early breast cancer (D-CARE): an international, multicentre, randomised, controlled, phase 3 trial. Lancet Oncol. 2020 Jan;21(1):60-72. doi: 10.1016/S1470-2045(19)30687-4. Epub 2019 Dec 2. PMID 31806543
- [Background] Coleman R, Zhou Y, Jandial D, Cadieux B, Chan A. Bone Health Outcomes from the International, Multicenter, Randomized, Phase 3, Placebo-Controlled D-CARE Study Assessing Adjuvant Denosumab in Early Breast Cancer. Adv Ther. 2021 Aug;38(8):4569-4580. doi: 10.1007/s12325-021-01812-9. Epub 2021 Jun 29. PMID 34185259
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 407 centers in Australia, Western Europe, Eastern Europe, Israel, North America, Asia, South America, South Africa, and Turkey from 02 June 2010 to 24 August 2012.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to 1 of 2 groups. Randomization was stratified based on breast cancer therapy/lymph node (LN) status, hormone receptor status, human epidermal growth factor receptor 2 (HER-2) status, age, and geographic region.
Groups:
- Placebo: Participants were randomized to receive placebo subcutaneous injections once every 3 or 4 weeks for approximately 6 months followed by placebo subcutaneous injections once every 3 months for 4.5 years.
- Denosumab: Participants were randomized to receive denosumab 120 mg subcutaneous injections once every 3 or 4 weeks for approximately 6 months followed by denosumab 120 mg subcutaneous injections once every 3 months for 4.5 years.
Period: Overall Study
Arm/Group | Placebo | Denosumab
Started | 2253 | 2256
Received Study Drug | 2229 | 2230
Completed | 27 | 28
Not Completed | 2226 | 2228
Not completed — Protocol-specified Criteria: Study Ended | 1524 | 1514
Not completed — Withdrawal by Subject | 369 | 385
Not completed — Death | 215 | 214
Not completed — Lost to Follow-up | 43 | 35
Not completed — Noncompliance | 22 | 20
Not completed — Disease Progression | 18 | 20
Not completed — Ineligibility Determined | 10 | 14
Not completed — Other | 14 | 11
Not completed — Adverse Event | 9 | 9
Not completed — Administrative Decision | 1 | 6
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab | Total
Number analyzed (Participants) | 2253 | 2256 | 4509
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.6) | 51.4 (10.7) | 51.5 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 1960 | 1959 | 3919
  65 - 74 years | 259 | 260 | 519
  75 - 84 years | 33 | 36 | 69
  ≥ 85 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2253 | 2256 | 4509
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1692 | 1676 | 3368
  Asian | 222 | 213 | 435
  Japanese | 134 | 135 | 269
  Hispanic/Latino | 112 | 135 | 247
  Black | 70 | 74 | 144
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 18 | 20 | 38
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 1165 | 1195 | 2360
  Postmenopausal | 1088 | 1061 | 2149
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 1913 | 1922 | 3835
    1 (Restricted but ambulatory) | 340 | 329 | 669
    2 (Ambulatory, unable to work) | 0 | 3 | 3
    Missing | 0 | 2 | 2
Breast Cancer Therapy / Lymph Node Status (Strata per Randomization) [Count of Participants; unit: Participants] — Breast cancer therapy / lymph node (LN) status:
  1. neo-adjuvant therapy / any LN status;
  2. adjuvant therapy / LN negative (based on axillary LN dissection, or based on sentinel node [SN] status);
  3. adjuvant therapy / LN positive
  Participants
    Neo-adjuvant therapy / any lymph node status | 550 | 552 | 1102
    Adjuvant therapy / lymph node negative | 68 | 65 | 133
    Adjuvant therapy / lymph node positive | 1635 | 1639 | 3274
Hormone Receptor Status (Strata per Randomization) [Count of Participants; unit: Participants] — Hormone receptor (estrogen receptor [ER] / progesterone receptor [PR]) status
  1. ER and/or PR positive
  2. ER and PR negative
  Participants
    ER and/or PR positive | 1740 | 1747 | 3487
    ER and PR negative | 513 | 509 | 1022
Human Epidermal Growth Factor Receptor 2 (HER-2) Status (Strata per Randomization) [Count of Participants; unit: Participants]
  HER-2 positive | 490 | 492 | 982
  HER-2 negative | 1763 | 1764 | 3527
Age (Strata per Randomization) [Count of Participants; unit: Participants]
  < 50 years | 1026 | 1029 | 2055
  ≥ 50 years | 1227 | 1227 | 2454
Geographic Region (Strata per Randomization) [Count of Participants; unit: Participants]
  Japan | 131 | 131 | 262
  Other | 2122 | 2125 | 4247
Molecular Subtypes of Breast Cancer [Count of Participants; unit: Participants] — Hormone receptor (HR; estrogen receptor [ER] / progesterone receptor [PR]); HR positive = ER and/or PR positive; HR negative = ER and PR negative
  Participants
    HR positive and HER-2 positive | 288 | 286 | 574
    HR positive and HER-2 negative | 1460 | 1458 | 2918
    HR negative and HER-2 positive | 163 | 168 | 331
    HR negative and HER-2 negative | 341 | 343 | 684
    Missing | 1 | 1 | 2
Lymph Node Status [Count of Participants; unit: Participants] — Clinical and pathologic regional lymph node (LN) status (by American Joint Committee on Cancer (AJCC)): N0 = no LN metastasis or pathologic (p) micrometastases <2.0 mm; N1 = Ipsilateral level I, II axillary (Ax) LN or p micrometastases >2.0mm or in internal mammary (IM) LN; N2 = fixed ipsilateral level I, II Ax LNs or clinically detected IM LNs only or pLN metastases in 4-9 Ax LNs; N3 = ipsilateral level III infraclavicular (IC) LNs or clinically detected IM LNs with other level I/II Ax LNs or supraclavicular (SC) LNs or pLN metastases in ≥10 Ax LNs; NX =LNs cannot be assessed.
  Participants
    N0 | 130 | 131 | 261
    N1 | 1369 | 1381 | 2750
    N2 | 506 | 505 | 1011
    N3 | 230 | 224 | 454
    Nx | 18 | 15 | 33
Breast Cancer Histopathologic Grade [Count of Participants; unit: Participants] — Tumor grade was determined according to the Nottingham Combined Histological Grading System, based on morphological features (tubule formation, nuclear pleomorphism, and mitotic count), by assigning a value of 1 (favorable) to 3 (unfavorable) for each feature. Scores for the 3 categories were added to give a combined histopathologic grade score: Grade (G)1 (low grade; favorable) = total score of 3, 4, or 5; G2 (intermediate) = total score of 6 or 7; G3 (high; unfavorable) = total score of 8 or 9.
  Participants
    Grade 1 = Low | 222 | 209 | 431
    Grade 2 = Intermediate | 1015 | 1079 | 2094
    Grade 3 = High | 938 | 906 | 1844
    Not Evaluable/Missing | 78 | 62 | 140

OUTCOME MEASURES:

1. Primary Outcome: Bone Metastasis-free Survival (BMFS)
Description: BMFS time was defined as the time interval from the randomization date to the first occurrence of bone metastasis or death from any cause, whichever came first. Participants last known to be alive with no bone metastasis were censored at their last assessment date, or at the primary analysis data cut-off date, whichever was first. Participants who had first occurrence of bone metastasis before randomization were censored at their randomization date.
  Bone metastasis must have been confirmed by central imaging analysis or by biopsy, Evidence of disseminated tumor cells in bone marrow was not sufficient for determination of disease recurrence. Development of new primary malignancy in bone was not considered as bone metastasis.
  Since the median BMSF time could not be estimated due to low number of events, the percentage of participants with an event (i.e., bone metastasis or death) is reported.
Time Frame: From randomization until the primary analysis data cut-off date of 31 August 2017; median (minimum, maximum) time on study was 67.2 (0.0, 85.9) and 67.0 (0.0, 86.6) months in each treatment group respectively.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 2253 | 2256
percentage of participants | 13.5 [12.1 to 15.0] | 12.9 [11.6 to 14.3]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.70, Stratified Log Rank; Stratified by breast cancer therapy/LN status, hormone receptor status, HER-2 status, age, and geographic region; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.82 to 1.14] — Based on a Cox proportional hazards model stratified by the randomization stratification factors; a hazard ratio < 1 favors denosumab

2. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS time was defined as the time interval from the randomization date to the date of first observation of disease recurrence or death from any cause, whichever was first. Participants last known to be alive with no disease recurrence were censored at their last assessment date, or at the primary analysis data cut-off date, whichever was first. Participants who had first disease recurrence before randomization were censored at their randomization date.
  Disease recurrence includes bone metastasis and extraosseous disease (EOD) confirmed by central imaging analysis or by biopsy/cytology. Development of non-breast cancer new primary malignancy was not considered as disease recurrence.
  Since the median DFS time could not be estimated due to low number of events, the percentage of participants with an event (i.e., disease recurrence or death) is reported.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 2253 | 2256
percentage of participants | 19.2 [17.6 to 20.8] | 19.6 [18.0 to 21.2]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.57, Stratified Log Rank; Stratified by breast cancer therapy/LN status, hormone receptor status, HER-2 status, age, and geographic region; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.91 to 1.19] — Based on a Cox proportional hazards model stratified by the randomization stratification factors; a hzard ratio < 1 favors denosumab

3. Secondary Outcome: Disease-free Survival (DFS) in the Postmenopausal Subset
Description: DFS time was defined as the time interval from the randomization date to the date of first observation of disease recurrence or death from any cause, whichever was first. Participants last known to be alive with no disease recurrence were censored at their last assessment date, or at the primary analysis data cut-off date, whichever was first. Participants who had first disease recurrence before randomization were censored at their randomization date.
  Disease recurrence includes bone metastasis and extraosseous disease (EOD) confirmed by central imaging analysis or by biopsy/cytology. Development of non-breast cancer new primary malignancy was not considered as disease recurrence.
  Since the median DFS time in the postmenopausal subset could not be estimated due to low number of events, the percentage of participants with an event (i.e., disease recurrence or death) is reported.
Time Frame: as for outcome 1
Population: Randomized participants postmenopausal at enrollment, defined as:
  * Undergone bilateral oophorectomy
  * Age ≥ 60 years
  * Age 45 to 59 years with 1 of the criteria, ie, either amenorrhea > 12 months with an intact uterus and ≥ 1 intact ovary; or amenorrhea for ≤ 12 months and follicle-stimulating hormone and estradiol in postmenopausal range.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 1088 | 1061
percentage of participants | 18.6 [16.3 to 20.9] | 20.3 [17.8 to 22.7]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.26, Stratified Log Rank; Stratified by breast cancer therapy/LN status, hormone receptor status, HER-2 status, age, and geographic region; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.92 to 1.36] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) time was defined as the time interval from the randomization date to the date of death from any cause. Participants last known to be alive were censored at their last contact date.
  Since the median time to overall survival could not be estimated at the time of the final analysis due to low numbers of events, the percentage of participants with an event (i.e., death) is reported.
Time Frame: From randomization until the end of study; median (minimum, maximum) time on study was 72.7 (0, 92) and 72.3 (0, 92) months in each treatment group respectively.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 2253 | 2256
percentage of participants | 9.5 [8.3 to 10.8] | 9.5 [8.3 to 10.7]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.94, Stratified Log Rank; Stratified by breast cancer therapy/LN status, hormone receptor status, HER-2 status, age, and geographic region; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.83 to 1.22] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Distant Recurrence-free Survival
Description: Distant recurrence-free survival (DRFS) was defined as the time interval from the randomization date to the date of first observation of distant disease recurrence or death from any cause, whichever came first. Participants last known to be alive, who had not experienced distant disease recurrence, were censored at their last assessment date, or at the primary analysis data cut-off date, whichever was first. Participants who had first distant recurrence before randomization were censored at their randomization date.
  Distant disease recurrence includes confirmed bone metastasis and extraosseous disease other than local-regional disease recurrence. Development of non-breast cancer new primary malignancy was not considered as distant disease recurrence.
  Since the median time to DRFS could not be estimated due to the low number of events, the percentage of participants with an event (i.e., distant recurrence or death) is reported.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 2253 | 2256
percentage of participants | 18.0 [16.4 to 19.6] | 18.7 [17.1 to 20.3]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.41, Stratified Log Rank; Stratified by breast cancer therapy/LN status, hormone receptor status, HER-2 status, age, and geographic region; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.92 to 1.21] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality includes deaths from first dose of study drug to the end of study date; median (min, max) time on study was 72.7 (0, 92) and 72.3 (0, 92) months for Placebo/Denosumab respectively. Adverse Events are from first dose of study drug to 30 days after last dose; median (min, max) time on treatment was 59.4 (0.7, 67) and 59.3 (0.7, 67) months for Placebo/Denosumab respectively.
Description: Eleven participants randomized to the placebo group received at least 1 dose of denosumab during the study and are counted in the denosumab group for safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo: Participants received placebo subcutaneous injections once every 3 or 4 weeks for approximately 6 months followed by placebo subcutaneous injections once every 3 months for 4.5 years.
- Denosumab: Participants received denosumab 120 mg subcutaneous injections once every 3 or 4 weeks for approximately 6 months followed by denosumab 120 mg subcutaneous injections once every 3 months for 4.5 years.
Arm/Group | Placebo | Denosumab
All-Cause Mortality (participants affected / at risk) | 215/2218 | 215/2241
Serious Adverse Events (participants affected / at risk) | 675/2218 | 702/2241
Other Adverse Events (participants affected / at risk) | 2123/2218 | 2149/2241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2218) | Denosumab (N=2241)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 17
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 114 | 83
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 36 | 35
Pancytopenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 4
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Metabolic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 2
Palpitations (Cardiac disorders) | 1 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
External ear disorder (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 5
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Thyroiditis acute (Endocrine disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 5 | 5
Diplopia (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinopathy proliferative (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Vitreous haematoma (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 6
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 1
Anal prolapse (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 4
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 15
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 2 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 10 | 18
Necrotising colitis (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 24
Adverse drug reaction (General disorders) | 1 | 0
Application site pain (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 3
BRCA2 gene mutation (General disorders) | 0 | 1
Breast complication associated with device (General disorders) | 1 | 0
Capsular contracture associated with breast implant (General disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 2
Chest pain (General disorders) | 6 | 5
Chills (General disorders) | 2 | 0
Complication associated with device (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 4
General physical health deterioration (General disorders) | 3 | 3
Generalised oedema (General disorders) | 0 | 1
Granuloma (General disorders) | 0 | 1
Idiosyncratic drug reaction (General disorders) | 0 | 1
Impaired healing (General disorders) | 3 | 0
Incarcerated hernia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 2
Infusion site extravasation (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 7
Mucosal inflammation (General disorders) | 4 | 2
Non-cardiac chest pain (General disorders) | 4 | 6
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 1 | 2
Peripheral swelling (General disorders) | 0 | 1
Pseudocyst (General disorders) | 0 | 1
Pyrexia (General disorders) | 33 | 37
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 6
Cholecystitis acute (Hepatobiliary disorders) | 4 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 5
Cholestasis (Hepatobiliary disorders) | 1 | 0
Gallbladder non-functioning (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Allergy to vaccine (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 2
Hypersensitivity (Immune system disorders) | 2 | 3
Reaction to preservatives (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 2 | 2
Appendiceal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 7
Appendicitis perforated (Infections and infestations) | 0 | 2
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Bacterial sepsis (Infections and infestations) | 1 | 2
Bartholinitis (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 3 | 5
Breast cellulitis (Infections and infestations) | 18 | 20
Bronchitis (Infections and infestations) | 3 | 4
Bursitis infective (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 3
Catheter site infection (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 30 | 34
Cellulitis staphylococcal (Infections and infestations) | 2 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 3
Clostridium difficile infection (Infections and infestations) | 2 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 2 | 1
Dengue fever (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 10 | 3
Device related sepsis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 8 | 1
Erysipelas (Infections and infestations) | 4 | 14
Erysipelothrix infection (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 4
Febrile infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Genital herpes simplex (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 4
Infected fistula (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 2 | 1
Infectious colitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 5 | 1
Intervertebral discitis (Infections and infestations) | 0 | 2
Labyrinthitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 6
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 3 | 2
Mastitis (Infections and infestations) | 8 | 12
Mastitis bacterial (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1
Mycobacterial infection (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 2 | 1
Neutropenic sepsis (Infections and infestations) | 14 | 15
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 3
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 1
Pericoronitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 1 | 0
Periumbilical abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 30 | 27
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 2
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 9 | 7
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 5
Pyelonephritis acute (Infections and infestations) | 1 | 4
Respiratory tract infection (Infections and infestations) | 1 | 3
Sebaceous gland infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 3
Septic shock (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 3
Skin infection (Infections and infestations) | 2 | 1
Staphylococcal infection (Infections and infestations) | 2 | 4
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 7
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 13 | 6
Urinary tract infection bacterial (Infections and infestations) | 2 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 3 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 1
Wound infection bacterial (Infections and infestations) | 3 | 6
Wound infection staphylococcal (Infections and infestations) | 3 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Exposure to radiation (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 6 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 2
Postmastectomy lymphoedema syndrome (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation mastitis (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 6 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 6 | 5
Skin flap necrosis (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 4 | 1
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Body temperature increased (Investigations) | 2 | 2
Bone scan abnormal (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 0 | 2
Neutrophil count abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2
Oestradiol increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Stroke volume increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 8 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 6
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Benign neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 15
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Retro-orbital neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 3
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral disorder (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 3 | 1
Cerebrospinal fistula (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 6 | 5
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Coma hepatic (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 4 | 3
Dystonia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 2
Facial neuralgia (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 10
Hemiparesis (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 3
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 4 | 5
Somnolence (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 9 | 2
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 3
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device expulsion (Product Issues) | 0 | 1
Device failure (Product Issues) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 7
Anxiety disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 8
Hypomania (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 2 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 6
Bladder perforation (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1
Breast haematoma (Reproductive system and breast disorders) | 1 | 2
Breast inflammation (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Breast necrosis (Reproductive system and breast disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 3
Cystocele (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 4 | 7
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 7 | 3
Ovarian enlargement (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 2 | 3
Uterine prolapse (Reproductive system and breast disorders) | 4 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20 | 17
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Segmented hyalinising vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Ankle arthroplasty (Surgical and medical procedures) | 0 | 1
Breast conserving surgery (Surgical and medical procedures) | 1 | 0
Breast operation (Surgical and medical procedures) | 1 | 0
Breast reconstruction (Surgical and medical procedures) | 2 | 2
Cancer surgery (Surgical and medical procedures) | 0 | 1
Catheter removal (Surgical and medical procedures) | 1 | 0
Cervical polypectomy (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 1
Mammoplasty (Surgical and medical procedures) | 1 | 0
Oophorectomy bilateral (Surgical and medical procedures) | 1 | 0
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1 | 0
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 1 | 0
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 12 | 9
Embolism (Vascular disorders) | 1 | 1
Embolism arterial (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 7
Intermittent claudication (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 2 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 2 | 0
Shock (Vascular disorders) | 1 | 0
Subclavian artery thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 3
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 3 | 0
Thrombosis (Vascular disorders) | 2 | 2
Varicose vein (Vascular disorders) | 1 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Cystitis escherichia (Infections and infestations) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Mastectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2218) | Denosumab (N=2241)
Anaemia (Blood and lymphatic system disorders) | 349 | 354
Leukopenia (Blood and lymphatic system disorders) | 154 | 145
Neutropenia (Blood and lymphatic system disorders) | 461 | 441
Lacrimation increased (Eye disorders) | 243 | 195
Abdominal pain (Gastrointestinal disorders) | 242 | 232
Abdominal pain upper (Gastrointestinal disorders) | 199 | 179
Constipation (Gastrointestinal disorders) | 635 | 626
Diarrhoea (Gastrointestinal disorders) | 638 | 660
Dyspepsia (Gastrointestinal disorders) | 245 | 273
Nausea (Gastrointestinal disorders) | 1095 | 1145
Stomatitis (Gastrointestinal disorders) | 398 | 399
Toothache (Gastrointestinal disorders) | 159 | 198
Vomiting (Gastrointestinal disorders) | 536 | 536
Asthenia (General disorders) | 404 | 407
Fatigue (General disorders) | 893 | 901
Influenza like illness (General disorders) | 145 | 154
Mucosal inflammation (General disorders) | 278 | 281
Oedema (General disorders) | 112 | 106
Oedema peripheral (General disorders) | 397 | 380
Pain (General disorders) | 178 | 156
Pyrexia (General disorders) | 342 | 338
Bronchitis (Infections and infestations) | 112 | 86
Influenza (Infections and infestations) | 117 | 117
Nasopharyngitis (Infections and infestations) | 290 | 292
Sinusitis (Infections and infestations) | 101 | 113
Upper respiratory tract infection (Infections and infestations) | 195 | 206
Urinary tract infection (Infections and infestations) | 149 | 177
Procedural pain (Injury, poisoning and procedural complications) | 161 | 170
Radiation skin injury (Injury, poisoning and procedural complications) | 351 | 361
Weight increased (Investigations) | 151 | 167
Decreased appetite (Metabolism and nutrition disorders) | 289 | 330
Hypocalcaemia (Metabolism and nutrition disorders) | 73 | 135
Arthralgia (Musculoskeletal and connective tissue disorders) | 974 | 973
Back pain (Musculoskeletal and connective tissue disorders) | 486 | 563
Bone pain (Musculoskeletal and connective tissue disorders) | 256 | 288
Muscle spasms (Musculoskeletal and connective tissue disorders) | 204 | 201
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 143 | 129
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 308 | 337
Myalgia (Musculoskeletal and connective tissue disorders) | 539 | 553
Neck pain (Musculoskeletal and connective tissue disorders) | 112 | 106
Pain in extremity (Musculoskeletal and connective tissue disorders) | 545 | 570
Pain in jaw (Musculoskeletal and connective tissue disorders) | 124 | 150
Dizziness (Nervous system disorders) | 255 | 273
Dysgeusia (Nervous system disorders) | 344 | 351
Headache (Nervous system disorders) | 567 | 527
Hypoaesthesia (Nervous system disorders) | 112 | 112
Neuropathy peripheral (Nervous system disorders) | 421 | 417
Paraesthesia (Nervous system disorders) | 197 | 216
Peripheral sensory neuropathy (Nervous system disorders) | 177 | 198
Anxiety (Psychiatric disorders) | 207 | 220
Depression (Psychiatric disorders) | 202 | 195
Insomnia (Psychiatric disorders) | 432 | 429
Breast pain (Reproductive system and breast disorders) | 189 | 178
Cough (Respiratory, thoracic and mediastinal disorders) | 426 | 410
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 268 | 280
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 151 | 168
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 176 | 157
Alopecia (Skin and subcutaneous tissue disorders) | 923 | 938
Dermatitis (Skin and subcutaneous tissue disorders) | 112 | 107
Dry skin (Skin and subcutaneous tissue disorders) | 133 | 125
Erythema (Skin and subcutaneous tissue disorders) | 226 | 260
Nail disorder (Skin and subcutaneous tissue disorders) | 264 | 275
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 114 | 138
Pruritus (Skin and subcutaneous tissue disorders) | 181 | 144
Rash (Skin and subcutaneous tissue disorders) | 372 | 392
Hot flush (Vascular disorders) | 645 | 669
Hypertension (Vascular disorders) | 209 | 195
Lymphoedema (Vascular disorders) | 350 | 392

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (3):
  • Study Protocol (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01077154/Prot_000.pdf
  • Statistical Analysis Plan: SAP 3.0 (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT01077154/SAP_001.pdf
  • Statistical Analysis Plan: SAP 3.0 Addendum (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT01077154/SAP_002.pdf